CLINICAL TRIAL: NCT05711251
Title: The Effect of the 10-week "Physical Activity in Health Promotion" Course on the Physical Activity Habits of University Students.
Brief Title: Physical Activity in Health Promotion Course on the Physical Activity Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AhiE
Record Dates: First submitted 2023-01-12; First posted 2023-02-02 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Physical Inactivity
Keywords: Physical Activity; University Students; Physical Activity Habit
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity in Health Promotion Group (Experimental): Students who chose the "Physical Activity in Health Promotion" course were included in the experimental group. The participants in this group took the courses shown in the weekly schedule below during the semester.
  1. Historical Development of Physical Activity
  2. Physical Activity Definition and Types
  3. Physical Activity Measurement
  4. Physical Fitness and Inactivity
  5. Physical Activity in Healthy Adults
  6. Physical Activity in Children
  7. Physical Activity in the Elderly
  8. Physical Activity for the Disabled
  9. Physical Activity at Work-I
  10. Physical Activity at Work-II
  Interventions: Other: Physical Activity in Health Promotion
- Control Group (No Intervention): Students who chose the "Posture Disorders" and "Waist and Neck Health" courses given by different instructors at the same time and day were included in the control group. the participants in this group took 2 different courses, shown in the weekly schedule below, at the same time, from different physiotherapists during the semester.
  Waist and Neck Health
  1. Functional anatomy, biomechanics and pathomechanics of the spine
  2. Risk factors for low back and neck pain
  3. Back and neck pain related disorders
  4. Outcome measures in low back and neck pain
  5. Treatment approaches
  6. Cervical and Lumbar disc lesions and physiotherapy
  7. Exercise principles for low back and neck pain
  8. Core stabilization, strengthening and stretching exercises
  9. Neck school: Organization, methods and principles
  10. Ergonomics

INTERVENTIONS:
Other: Physical Activity in Health Promotion — During the term, the participants in the study group took lessons on many subjects, from the benefits of physical activity to suggestions to increase physical activity at work and in daily life.
  Arms: Physical Activity in Health Promotion Group

SUMMARY:
The goal of this interventional study is to learn about 10-week "Physical Activity in Health Promotion" course on the physical activity habits of university students. The main question it aims to answer are:

• What is the effect of 10-week "Physical Activity in Health Promotion" course on the physical activity habits of university students in Ahi Evran University.

Healthy participants will take elective courses named:

* Physical Activity in Health Promotion
* Waist and Neck Health
* Posture Disorders

DETAILED DESCRIPTION:
A healthy lifestyle must include physical activity, especially for university students. There is now substantial data supporting the numerous physical, psychological, aesthetic, and social advantages of frequent engagement in physical activities. A number of illnesses and ailments, such as coronary artery disease, heart disease, stroke, diabetes, high blood pressure, colon cancer, breast cancer, and overweight and obesity are all made less likely by regular physical activity. Numerous research in the area have documented a tendency toward less physical activity among adults, adolescents, and children in various civilizations. The level of physical activity among university students was found to be relatively low during the pandemic, and this process also had a detrimental impact on the students' levels of depression and quality of life. Walking, moderate, vigorous, and overall physical activity levels have decreased among university students from many nations who have been quarantined due to the COVID-19 epidemic.

One of the most popular teaching methods in medical school is the lecture course, which has the benefit of allowing for the dissemination of knowledge to a large number of students and has the potential to be effective in conveying factual information. Whether or not it is successful, lecturing is still the most popular teaching style since it is affordable and useful, especially when there are many students and few resources. Physical education provides cognitive content and instruction designed to develop motor skills, knowledge, and behaviors for physical activity and physical fitness. Supporting schools to establish physical education can provide students with the ability and confidence to be physically active for a lifetime. However, the number of studies investigating the effects of physical activity classes or physical activity education on students' physical activity habits is very low in the literature.

The "Physical activity for the health promotion" course given at Ahi Evran University was added to the curriculum in order to increase the physical activity knowledge and levels of university students. The course was a common elective course open to all university students except the physiotherapy and rehabilitation department. The aim of this study is to investigate the effect of the "Physical Activity in Health Promotion" course on the physical activity levels of university students. For this purpose, our hypothesis is: "Physical activity for the promotion of health" course will change the physical activity habits of university students.

ELIGIBILITY:
Inclusion Criteria:

* Healthy students who took elective courses

Exclusion Criteria:

* To be involved in another study,
* Having a systemic disease that limits physical activity,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 10 weeks
  The IPAQ questionnaires list activities and request estimates of durations and frequencies for each activity engaged in over the past week. Durations are multiplied by known METs per activity and the results for all items are summed for the overall physical activity score. Scores for walking and for moderate and vigorous activities are sums of corresponding item scores.
Domain-Specific Physical Activity Efficacy Questionnaire (DSPAEQ) | 10 weeks
  The DSPAEQ consists of 26 items and asks students how confident they are to engage in physical activity across five different domains [ambulatory (6 items), household (5 items), leisure-time (6 items), transportation (3 items), and school (6 items)]. Participants responded to each item using a 10-point scale ranging from 0% (not at all confident) to 100% (completely confident).

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared online with Google Drive
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: a year study finished
Access Criteria: With permission
URL: http://docs.google.com/spreadsheets/d/1MBgJUfi0PfeD20mf3npJtoLByeSAfzmtvjZz1YidkDc/edit?usp=sharing

REFERENCES:
- [Background] Alaagib NA, Musa OA, Saeed AM. Comparison of the effectiveness of lectures based on problems and traditional lectures in physiology teaching in Sudan. BMC Med Educ. 2019 Sep 23;19(1):365. doi: 10.1186/s12909-019-1799-0. PMID 31547817
- [Background] Lopez-Valenciano A, Suarez-Iglesias D, Sanchez-Lastra MA, Ayan C. Impact of COVID-19 Pandemic on University Students' Physical Activity Levels: An Early Systematic Review. Front Psychol. 2021 Jan 15;11:624567. doi: 10.3389/fpsyg.2020.624567. eCollection 2020. PMID 33519653